CLINICAL TRIAL: NCT03498872
Title: Exercise and the Brain in Health & Disease: The Added Value of Human-Centered Robotics
Brief Title: Strategic Research Program 17 (VUB Funding)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Prof. Dr., Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROJECT-ID SRP 17
Record Dates: First submitted 2018-04-03; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Prosthesis User; Amputation; Traumatic, Limb, Lower
Keywords: AMPfoot; Prosthetics; gait; electro-encephalography; dual-task walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Able-bodied individuals (Active Comparator)
  Interventions: Other: No intervention
- Transtibial amputee (Experimental)
  Interventions: Device: AMPfoot 4.0
- Transfemoral amputee (Experimental)
  Interventions: Device: AMPfoot 4.0

INTERVENTIONS:
Device: AMPfoot 4.0 — The novel prosthetic device, i.e. AMPfoot 4.0, was tested during walking in amputees. A dual-task was conducted and non-invasive electro-encephalography was used to investigate neural dynamics.
  Arms: Transfemoral amputee; Transtibial amputee
Other: No intervention — The control group included healthy subjects. Comparisons were made between amputees and able-bodied individuals.
  Arms: Able-bodied individuals

SUMMARY:
Objectives: The main objectives are to determine neural dynamics during gait using electro-encephalography as well as brain sources and to investigate the attentional demand during walking in able-bodied individuals, and individuals with an amputation.

Materials & Methods: 6 able-bodied individuals conducted one experimental trial, and 6 unilateral transtibial and 6 unilateral transfemoral amputees performed 2 experimental trials; the first with the current and the second with a novel powered transtibial prosthesis, i.e. the Ankle Mimicking Prosthetic foot 4.0. Each experimental trial comprised 2 walking tasks; 6 and 2min treadmill walking at normal speed interspersed by 5min of rest. During 6min walking the sustained attention to response (go-no go) task, with measures reaction time and accuracy, was performed. Electro-encephalographic (EEG) data were gathered when subjects walked 2min. Motor-related cortical potentials and brain activity during gait are extracted using EEG.

DETAILED DESCRIPTION:
Detailed description of the novel device:

The device mainly distinguishes itself from commercial prostheses thanks to its new type of actuation providing a compact and energy efficient solution to the challenge of ankle-foot actuation. This new actuation method consists of using springs, a servo motor and a locking mechanism, coupled with a sensory network providing intelligence to the robotic device. The AMPfoot 4.0 design is also based on previous research conducted on the AMP-Foot 2. However, it is important to note that in contrast with its preceding designs, the AMP-Foot 4.0 does not provide active propulsion at push-off.

During walking, the AMP-Foot 4.0 working principle is divided into two main logic sequences, i.e. the stance and the swing phase. These two phases are detected by analyzing gyroscope and acceleration measurements from an Inertial Measurement Unit chip. During the stance phase, the ankle performs a dorsi-flexing movement while a plantar-flexing torque is applied at the ankle. The person's gravitational potential energy is stored into elastic potential energy by means of the used spring. It is this spring that provides the plantar-flexing torque required at the ankle as reaction to the movement of the user. Due to the use of a locking system, the prosthesis can adapt its so-called zero torque rest point depending on the slope or stride length of the user. This provides adaptability and therefore greater comfort compared to prostheses with a fixed zero torque rest point. During the swing phase, the locking mechanism unlocks to free the ankle movement. Parallel springs external to the stance system are then activated to reset the foot to its initial position. From that moment, the device is ready for a new step.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral amputees
* Unilateral transtibial amputees
* Able-bodied individuals

Exclusion Criteria:

* Children
* Functional k-level lower than 4 (Amputee has the ability for prosthetic ambulation that exceeds basic ambulation skills, exhibiting high impact, stress or energy levels)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Reaction time (in ms) of responses during go - no go cognitive task | Through study completion, a period of 2 months
  Time between visual stimulus and motor response (pushing button)
Accuracy (in percentage) of correct responses during go - no go cognitive task | Through study completion, a period of 2 months
  Accuracy of motor responses to visual stimuli
EEG extracted brain signals, i.e. motor-related cortical potentials | Through study completion, a period of 2 months
  Non-invasive electro-encephalography was used to determine electro-cortical potentials and brain sources of these potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No